CLINICAL TRIAL: NCT01104597
Title: Assessment of Subclinical Atherosclerosis in Healthy Adult Immigrant Asian Indians Using Flow Mediated Endothelial Dysfunction Method
Brief Title: Study to Evaluate Subclinical Atherosclerosis (an Early Sign of Heart Disease) in Healthy Adult Immigrant Asian Indians
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were enrolled into the study
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Rajiv Jauhar, Chief, Cardiology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-272
Record Dates: First submitted 2010-04-09; First posted 2010-04-15 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy Asian Indians and Caucasians
MeSH Terms: interventions — Nitroglycerin; Administration, Sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Flow Mediated Doppler (FMD) — Non-invasive assessment of flow-mediated dilation (FMD) will be performed using brachial artery ultrasound.
Drug: Nitroglycerin 0.4 mg sublingual — Nitroglycerin 0.4 mg (a small tablet that dissolves under the tongue) will be given to dilate the arteries. Images of the arm will be recorded via non-invasive flow-mediated doppler for 5 minutes to assess for endothelium dysfunction. as outlined above.

SUMMARY:
Previous research has shown that Asian Indians are at relatively high risk for developing diabetes, heart problems and high blood pressure.

The purpose of this study is to evaluate subclinical atherosclerosis (an early sign of heart disease) which may be associated with abnormalities like diabetes mellitus, hypertension (high blood pressure), high cholesterol and heart problems.

Endothelium is the inner lining of your blood vessels. Endothelial dysfunction is found more in people with diabetes. In addition, high body mass index (BMI) is a strong risk factor for developing metabolic abnormalities like diabetes mellitus. This research study may provide information as to how useful endothelial dysfunction will be to detect people at risk of metabolic abnormalities and heart disease at an early stage.

Two groups of subjects will be enrolled. Caucasians and Asian Indians There will be a total of 100 subjects participating in this study. Approximately 50 Caucasians and 50 Asian Indians will be enrolled. Caucasians will serve as the control group for this study.

ELIGIBILITY:
Inclusion Criteria:

* Asian Indians and Caucasians between the ages of 20 and 65 living in the boroughs of New York City and the Long Island area.

Subjects must provide a record of blood results completed within the past year to determine eligibility (hematology and chemistry results).

Exclusion Criteria:

* Subjects with major underlying medical problems, including diabetes, hypertension, coronary artery disease (CAD), hyperlipidemia, systolic blood pressure below 90 mm Hg and liver or kidney disease will be excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assessment of subclinical atherosclerosis in healthy adult immigrant Asian Indians using flow mediated endothelial dysfunction method | April 2010 to April 2012
  To evaluate subclinical atherosclerosis (an early sign of heart disease) which may be associated with abnormalities like diabetes mellitus, hypertension (high blood pressure), high cholesterol and heart problems.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Jauhar, MD, Principal Investigator — Northwell Health